CLINICAL TRIAL: NCT01558141
Title: Follicular Flushing on Cycle Outcomes in Poor Responders
Brief Title: Follicular Flushing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1108011882
Record Dates: First submitted 2012-02-16; First posted 2012-03-20 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2015-06

CONDITIONS: Fertilization
Keywords: IVF stimulation.; Poor responders.; IVF patients with poor response to stimulation
MeSH Terms: interventions — Culture Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Follicular flushing (Active Comparator): Flushing follicles with embryo culture media prior to aspiration.
  Interventions: Other: Aspiration without flushing follicles with culture media; Other: Follicular Flushing

INTERVENTIONS:
Other: Aspiration without flushing follicles with culture media — Aspiration without flushing follicles with culture media.
Other: Follicular Flushing — Flushing follicles with embryo culture media prior to aspiration.

SUMMARY:
Patients with infertility often undergo in vitro fertilization (IVF) to achieve a pregnancy, which involves ovarian stimulation, monitoring of follicular growth, oocyte retrieval, sperm insemination, embryo culture and embryo transfer.

The oocytes are removed during surgery by aspirating the follicles using a single lumen needle with an ultrasound to guide the procedure. There is some data that flushing the follicles with embryo culture media before aspiration using a double lumen needle increases the number of oocytes retrieved, particularly among poor responding patients for whom each additional oocyte recovered may substantially alter the outcome of that IVF cycle.

The objective of the research is to evaluate the effect of follicular flushing in poor responders on IVF cycle outcomes.

DETAILED DESCRIPTION:
Patients with infertility often undergo in vitro fertilization (IVF) to achieve a pregnancy, which involves ovarian stimulation, monitoring of follicular growth, oocyte retrieval, sperm insemination, embryo culture and embryo transfer. The number of embryos obtained is dependent on the number of oocytes retrieved.

The objective of the research is to evaluate the effect of follicular flushing in poor responders on IVF cycle outcomes, including the number of oocytes retrieved, number of mature oocytes, fertilization rate, number of embryos transferred, implantation rate, miscarriage rate, live birth rate, operating room time, and luteal estradiol and progesterone levels.

The research entails a prospective, randomized, controlled trial of poor-responder patients who are undergoing IVF treatment at The Ronald O. Perelman and Claudia Cohen Center for Reproductive Medicine, defined as patients who have ≤ 4 follicles that are ≥ 12mm on the day of hCG trigger.

Patients identified as poor responders will be consented and randomized to follicular flushing versus aspiration without flushing. A 2-5mL flush using embryo culture media followed by aspiration of the follicle will be performed in the patients randomized to the flushing group, with subsequent flushes until an oocyte is identified or up to 4 flushes maximum.

Patients being enrolled in this research study will undergo IVF regardless of participation in this research study.

Randomization:

A series of randomized blocks of 2 will be generated for the study. This will provide assurance that after two patients are enrolled, there will be one patient assigned to each group- follicular flushing versus aspiration without flushing. This process of blocked randomization ensures an equal distribution between the two study arms of patients.

ELIGIBILITY:
Inclusion Criteria:

* Pts ages 18-45 undergoing IVF
* Pts with ≤ 4 follicles that are ≥ 12mm on day of HCG

Exclusion Criteria:

* Pts undergoing natural cycles (i.e. those with intentionally low # of follicles)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2011-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
FOLLICULAR FLUSHING ON CYCLE OUTCOMES IN POOR RESPONDERS | 2 weeks
  To evaluate the number of oocytes retrieved with follicular flushing in poor responders

SECONDARY OUTCOMES:
FOLLICULAR FLUSHING ON CYCLE OUTCOMES IN POOR RESPONDERS | 2 weeks
  To evaluate:
  - # of embryos transferred
FOLLICULAR FLUSHING ON CYCLE OUTCOMES IN POOR RESPONDERS | 2 weeks
  Fertilization rates.
FOLLICULAR FLUSHING ON CYCLE OUTCOMES IN POOR RESPONDERS | 2 weeks
  Implantation rates
FOLLICULAR FLUSHING ON CYCLE OUTCOMES IN POOR RESPONDERS | 2 weeks
  Pregnancy rates
FOLLICULAR FLUSHING ON CYCLE OUTCOMES IN POOR RESPONDERS | 2 weeks
  Live birth rates
FOLLICULAR FLUSHING ON CYCLE OUTCOMES IN POOR RESPONDERS | 2 weeks
  Operating room anesthesia time.
FOLLICULAR FLUSHING ON CYCLE OUTCOMES IN POOR RESPONDERS | 2 weeks
  Luteal E2 level.
FOLLICULAR FLUSHING ON CYCLE OUTCOMES IN POOR RESPONDERS | 2 weeks
  Luteal P4 level.

CONTACTS AND LOCATIONS:
Overall Officials: Steven D. Spandorfer, MD, Principal Investigator — Weill Medical College of Cornell
Locations (1):
- New York Presbyterian Hospital, New York, New York, United States

REFERENCES:
- [Derived] Mok-Lin E, Brauer AA, Schattman G, Zaninovic N, Rosenwaks Z, Spandorfer S. Follicular flushing and in vitro fertilization outcomes in the poorest responders: a randomized controlled trial. Hum Reprod. 2013 Nov;28(11):2990-5. doi: 10.1093/humrep/det350. Epub 2013 Sep 5. PMID 24014603